CLINICAL TRIAL: NCT03145532
Title: Transcranial Direct-Current Stimulation (tCDS) and Robotics for Children With Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blythedale Children's Hospital (Other)
Responsible Party: Principal Investigator, Kathleen Friel, Director, Cerebral Palsy Research, Blythedale Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-1003KF
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Hemiplegia
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Children will be randomized to receive either real or sham tDCS plus robotic training. Children in the sham group will be given the opportunity to repeat the protocol and receive real stimulation after they complete the sham protocol.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: tDCS will be blinded in that even children in the sham group will receive a low level of stimulation for a brief period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS plus robotic training (Experimental): Children will receive 20 min of real tDCS stimulation per session, followed by robotic training for 1 hr.
  Interventions: Other: tDCS plus robotic training
- Sham tDCS plus robotic training (Sham Comparator): Children will receive 20 min of sham tDCS stimulation per session, followed by robotic training for 1 hr.
  Interventions: Other: tDCS plus robotic training

INTERVENTIONS:
Other: tDCS plus robotic training — Children will first receive 20 min of tDCS (real or sham, see Arms), then will receive 1 hr of upper limb robotic therapy in which the child will use their impaired arm and hand to move a joystick controlling a cursor to a set of targets on a video screen in front of the child.

SUMMARY:
Hemiplegia occurs when the function of motor areas in the brain become impaired, predominantly unilaterally, during perinatal development. Children with hemiplegia show impairments in motor control of the affected side of the body. Impairments in use of the upper extremity are common, and lead to functional disability throughout the lifespan of a person with hemiplegia. Upper extremity impairments can severely affect a person's ability to carry out activities of daily living.

The goal of this study at Blythedale Children's Hospital is to test the efficacy of transcranial direct current stimulation (tDCS) and robotic upper extremity therapy in improving upper extremity function in children with unilateral cerebral palsy. This study will test the hypothesis that physical rehabilitation, provided by repetitive arm movements guided by a robot, will improve upper extremity function in children with hemiplegia, and that this improvement can be enhanced by transcranial direct current stimulation of motor cortex immediately before robotic training.

DETAILED DESCRIPTION:
This sham-controlled, double-blind study will be completed at Blythedale Children's Hospital.

Detailed procedures

Robotic Device and Patient Position

The investigators will use existing robots at Blythedale, which are FDA approved robotic devices that move the shoulder-and-elbow, or wrist-and-forearm, or the Typo Amadeo digit training robot.

All robots: The subject will sit in a foam-padded chair facing the robot and a video screen.

Planar (shoulder-elbow) and wrist robots: The arm will be abducted, forearm supported, and hand lightly grasping the robot handle, and velcro straps will lightly hold the forearm and fingers secure. A cursor on the video screen will display the targets and track the movement of the patient's arm.

Amadeo: The arm will be abducted, forearm supported, and digits attached to the robot with magnets. Velcro straps will lightly hold the forearm and fingers secure. A cursor on the video screen will display the targets and track the movement of the patient's fingers.

Robotic Training

Participants will receive a total of 12 sessions comprising 1 hour of interactive robotic training. Participants will have two to four study visits per week. During one visit, the child will receive tDCS + 1 hr training on the shoulder-elbow MIT Manus robot, and on the second visit of the week, the child will receive tDCS + 1 hr training on the wrist MIT Manus robot.

The interactive robot features involve visuomotor tasks, moving the robotic manipulandum according to targets on a computer screen mounted at eye level. A key feature of MIT robots is the low near isotropic inertia and reduced friction in the robot arm so that, when appropriate, it can "get out of the way." The force required to move the robotic arm is minimal, comparable to moving unrestricted, and if a patient cannot move the robot arm, it will guide the limb to provide an adaptive sensorimotor experience.

Transcranial Direct Current Stimulation

A current up to 1.5mA current will be delivered using surface rubber-carbon electrodes (35cm2) with surrounding saline soaked sponges (0.9% NaCl) by a battery driven, constant current stimulator (maximum output 2mA). Participants will receive stimulation for 20 minutes while seated (before robotic motor training), with the anode over the optimal site for first dorsal interosseous (FDI) as identified using TMS, and the cathode on the contralateral supraorbital area. Sham tDCS: comparable set-up to real tDCS, 30 sec real current ramping to current up to 1.5mA at commencement, then after 5 sec a slow decrease but to no current sustained for 20mins.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17
* Participant and caregiver willing and able to provide informed consen/assent
* Diagnosis of hemiplegia
* Joint mobility: wrist extension, 20º, metacarpophalangeal and proximal interphalangeal joints 10º

Exclusion Criteria:

* Cognitive deficits that impede understanding of study protocol
* Current medical illness unrelated to CP
* Visual problems (uncorrected by glasses/contact lenses)
* High motor ability in affected arm Pre-intervention screening measures; Motor activity log, score > 2.5 ( > slight-to-moderate)
* Severe spasticity Pre-intervention screening measures; Modified Ashworth test, score > 3 ( > moderate)
* Lack of asymmetry in hand function
* Orthopedic surgery in affected arm within 2 years
* Dorsal root rhizotomy
* Botulinum toxin therapy in either upper extremity during last 2 months, or planned during study period
* Currently receiving intrathecal baclofen
* Seizure beyond age 2, use of anti-seizure medication, history of epilepsy (in self or first degree relatives), brain surgery, cranial metal implants, structural brain lesion, devices that may be affected by TMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* True positive response on the Transcranial Magnetic Stimulation Safety Screen
* Current use of medications known to lower the seizure threshold
* Previous episode of neurocardiogenic syncopy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment after intervention | Within one week after the intervention ends
  Assessment of how well children incorporate both hands into bimanual task performance, using an assessment tool called the "Assisting Hand Assessment"
Change in Jebsen-Taylor Test of Hand Function after intervention | Within one week after the intervention ends
  Assessment of unimanual movement speed
Change in Box and blocks test after intervention | Within one week after the intervention ends
  Assessment of unimanual function

CONTACTS AND LOCATIONS:
Locations (1):
- Kathleen Friel, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share deidentified data in the NIH DASH (Data and Specimen Hub) database, sponsored by the National Institute of Child Health and Development (NICHD). Data will be archived to DASH upon study completion.